CLINICAL TRIAL: NCT06099249
Title: Validation of ECG Measurement and Atrial Fibrillation Detection Function of ASUS ECG App
Brief Title: Validation of ECG Measurement and Atrial Fibrillation Detection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: ASUSTek Computer INC. (Industry)
Collaborators: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Validation of ECG Measurement
Record Dates: First submitted 2023-10-16; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation
Keywords: Cardiovascular diseases; Heart Diseases; Arrhythmia; Cardiac
MeSH Terms: conditions — Atrial Fibrillation; Cardiovascular Diseases; Heart Diseases; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No_AFib_Group: Subjects enrolled into No_AFib_Group must have no known medical history of AFib and in normal sinus rhythm at the time of screening.
  Interventions: Device: ASUS ECG App
- AFib_Group: Subjects enrolled into AFib_Group must have a known diagnosis of persistent or permanent AFib and be in AFib at the time of screening.
  Interventions: Device: ASUS ECG App

INTERVENTIONS:
Device: ASUS ECG App — The procedure will commence with instructing the participants to become acquainted with the ASUS ECG App. Following this introduction, participants will be asked to sit quietly for a 5-minute resting period before undergoing a 12-lead ECG recording, which will last for approximately 30 seconds. The participant will be guided to simultaneously record a separate single-lead ECG using the ASUS ECG App. Both data streams will be synced together by the Study Staff. Each participant will undergo a total of three trials involving the simultaneous recording of a 12-lead ECG and a single-lead ECG using the ASUS ECG App.

SUMMARY:
Atrial fibrillation (AFib) is a common type of cardiac arrhythmia in clinical practice, affecting millions of people worldwide. Early detection and treatment of atrial fibrillation are crucial in preventing serious complications such as stroke and heart failure. In recent years, with the flourishing development of wearable devices and mobile technology, electrocardiogram (ECG) measurement applications embedded in smartwatches have gradually become a non-invasive and convenient method for heart rate monitoring. However, the accuracy of these devices has not yet been fully determined. This study aims to verify the ECG measurement and atrial fibrillation detection function of the ASUS ECG App. The accuracy of the ECG application in detecting atrial fibrillation and measuring ECG will be evaluated by comparison with standard 12-lead ECGs.

DETAILED DESCRIPTION:
This study plans to recruit 602 adults over the age of 18. All participants will undergo heart rate measurements using both the smartwatch ECG application and the 12-lead ECG. The heart rate measurement using the ECG application will be operated by the participants themselves under the guidance of the testing personnel. The 12-lead ECG will be operated by trained medical professionals. The results of the heart rate measurement from both devices will be recorded synchronously, and the consistency of heart rate interpretation and ECG waveforms between the smartwatch ECG application and the 12-lead ECG measurement will be compared to verify the accuracy of the ECG application.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to participate in the study procedures as described in the consent form
* Able to communicate effectively with and follow instructions from the study staff
* Subjects enrolled into No_AFib_Group must have no known medical history of AFib and in normal sinus rhythm at the time of screening.
* Subjects enrolled into AFib_Group must have a known diagnosis of persistent or permanent AFib and be in AFib at the time of screening.

Exclusion Criteria:

* Physical disability that precludes safe and adequate testing.
* Mental impairment as determined by the Investigator.
* Pregnant women at the time of the screening visit.
* Subjects with any Medical History, Physical exam, vital sign or any other study procedure finding/assessment that in the opinion of the investigator could compromise subject safety during study participation or interfere with the study integrity and/or the accurate assessment of the study objectives. This includes patients with known untreated medical conditions that are considered clinically significant by the Investigator, such as but not limited to significant anemia, important electrolyte imbalance and untreated or uncontrolled thyroid disease.
* Physical exam limitations include but not limited to open wound(s) on the wrist and forearm where the subject will be wearing the watch.
* Any history of wrist surgery with scarring in the area of the sensor location on the wrist where the subject will be wearing the watch.
* Vital signs measurement, medical history, or physical exam finding that makes the subject inappropriate for participation according to the Investigator.
* Tattoos or moles in the area of the sensor location on the wrist where the subject will be wearing the watch.
* Skin conditions on either wrist that would preclude subject from wearing watch on either wrist. Severe symptomatic(or active) overly dry/injured skin, skin disorders, or allergic skin reactions such as eczema, rosacea, impetigo,dermatomyositis or allergic contact dermatitis on wrist and locations where the electrodes will be placed (e.g.

chest,forearms, stomach), as determined by the investigator.

* Known allergy or significant sensitivity to medical adhesives, isopropyl alcohol, or ECG patch.
* Clinically significant hand tremors as judged by the Investigator.
* Subjects with implanted cardiac devices such as a Pacemaker or an automated Implantable Cardioverter-Defibrillator.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include two cohorts of subjects:
  1. No_AFib_Group will include subjects with no known history of AFib and are in normal sinus rhythm at time of screening.
  2. AFib_Group will include subjects with known persistent or permanent or chronic AFib who are in AFib at the time ofscreening.
  The following age and gender enrollment targets will be adhered to during subject recruitment:
  1. A minimum of 20% of subjects in both cohorts will be enrolled in each of the age categories of 55 to 64, and ≥65years, and a minimum of 10% of subjects in both cohorts in the age category of <55 years.
  2. At least 40% of subjects in No_AFib_Group will be female. At least 20% of subjects in AFib_Group will be female.
Sampling Method: Non-Probability Sample
Enrollment: 602 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity | One day
  Sensitivity and specificity of the ASUS ECG App in detecting AFib compared with physician-adjudicated 12-lead ECG will be calculated.

SECONDARY OUTCOMES:
Equivalence of the ECG app waveform to Lead I from a 12-lead ECG | One day
  Equivalence of the ECG app waveform to Lead I from a 12-lead ECG as measured by acceptable morphology of PQRST complexes and R-Wave amplitude agreement

IPD SHARING:
Plan to Share IPD: No